CLINICAL TRIAL: NCT04802993
Title: Survival Among Elderly Patients in Sweden With Right-sided Pancreatic Adenocarcinoma Depending on Resection Rate of Pancreaticoduodenectomy
Brief Title: Survival Among Patients With Pancreatic Cancer Depending on Surgical Resection Rate
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Bergthor Björnsson, Ass. Professor, senior consultant, Linkoeping University
Other Study IDs: 2017/151-31
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- All patients with pancreatic ductal adenocarcinoma aged 70 years and older: All patients in the registry aged 70 years and older with right-sided pancreatic ductal adenocarcinoma
  Interventions: Other: Resection rates
- All patients with pancreatic ductal adenocarcinoma aged 70-79 years: All patients in the registry aged 70-79 years with right-sided pancreatic ductal adenocarcinoma
  Interventions: Other: Resection rates
- All patients with pancreatic ductal adenocarcinoma aged 80 years and older: All patients in the registry aged 80 years and older with right-sided pancreatic ductal adenocarcinoma
  Interventions: Other: Resection rates
- All patients resected with pancreaticoduodenectomy, all ages: All patients in the registry resected with pancreaticoduodenectomy during the study period
  Interventions: Other: Resection rates
- All patients resected with pancreaticoduodenectomy, aged 70-79 years: All patients in the registry resected with pancreaticoduodenectomy during the study period, aged 70-79 years
  Interventions: Other: Resection rates
- All patients resected with pancreaticoduodenectomy, aged 80 years and older: All patients in the registry resected with pancreaticoduodenectomy during the study period, aged 80 years and older
  Interventions: Other: Resection rates

INTERVENTIONS:
Other: Resection rates — All groups are divided into one high- and one low resection rate group depending on percentage of patients with pancreatic ductal adenocarcinoma resected per county and year (first three groups) and resection rate of pancreaticoduodenectomy per 100 000 inhabitants per county (last three groups)

SUMMARY:
The primary aim of this population-based study is to investigate how a high resection rate of pancreaticoduodenectomy affects overall survival among patients aged ≥70 years with pancreatic ductal adenocarcinoma. The secondary aim is to determine if a high resection rate of pancreaticoduodenectomy increases perioperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed between 1 January 2010 and 31 December 2018
* Registered in the Swedish National Registry for tumours in the pancreatic and periampullary region
* Either a diagnosis of pancreatic ductal adenocarcinoma of the pancreatic head or having been resected with pancreaticoduodenectomy

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients registered in the Swedish National Registry for tumours in the pancreatic and periampullary region diagnosed with right-sided pancreatic adenocarcinoma or resected with pancreaticoduodenectomy
Sampling Method: Non-Probability Sample
Enrollment: 5123 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | A little more than 10 years (from first patient to vital status)
  Overall survival among patients aged 70 years and over with pancreatic ductal adenocarcinoma in the pancreatic head

SECONDARY OUTCOMES:
Severe complications after pancreaticoduodenectomy | Around 10 years (patients diagnosed between 1 January 2010 and 31 December 2018, latest dismissal from hospital january 2020)
  The rate of severe complications among patients aged 70 years and over who had undergone pancreaticoduodenectomy for any reason

IPD SHARING:
Plan to Share IPD: No
The data cannot be further shared by the researchers but is available on application to the Swedish National Registry for tumours in the pancreatic and periampullary region, provided the application is approved by the Swedish Ethical Review Authority